CLINICAL TRIAL: NCT00521508
Title: Role of CD4+CD25+FoxP3+ Regulatory T Cells in Pathogenesis of Primary IgA Nephropathy
Brief Title: Role of Regulatory T Cells in Pathogenesis of Primary IgA Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Clément CAILLAUX, CHU Saint-Etienne
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0608118; 2007-A00129-44; DGS 2007-0184
Record Dates: First submitted 2007-08-27; First posted 2007-08-28 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Glomerulonephritis, IGA
Keywords: IgA; kidney; Berger'disease; regulatory T cells; pathogenesis of Berger's disease
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Transcription, Genetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Other): Patient affected by Berger's disease confirmed by renal biopsy with increased rate of Ig A
  Interventions: Procedure: gene transcription and cytometry
- 2 (Other): Patient affected by Berger's disease with normal rate of Ig A
  Interventions: Procedure: gene transcription and cytometry
- 3 (Other): Healthy volunteers
  Interventions: Procedure: gene transcription and cytometry

INTERVENTIONS:
Procedure: gene transcription and cytometry — samply of 30 ml of blood

SUMMARY:
Along structural IgA abnormalities, hyperproduction of IgA is thought to play a role in the pathogenesis of primary IgA nephropathy. CD4+CD25+Fox3P regulatory T cells are instrumental in suppressing adaptative immune responses, including B cells production of immunoglobulins. We, the researchers at Centre Hospitalier Universitaire de Saine Etienne, will test the hypothesis that IgA production in patients with IgA nephropathy is dysregulated because of a quantitative and/or qualitative defect of CD4+CD25+FoxP3+ regulatory T cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathogenesis of Berger's disease confirmed by renal biopsy
* Glomerular filtration > 60 ml/min/1,73m2
* Written informed consent
* Patient affiliated to social insurance

Exclusion Criteria:

* Immunosuppressor treatment within 6 months before the study inclusion
* Clinical infection within 2 months before the study inclusion
* C-reactive protein (CRP) > 10 mgL-1

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
proportion averages of cells CD4+CD25+CD127 low T in peripheral blood | inclusion

SECONDARY OUTCOMES:
average relative expression of genes FoxP3, CTLA4, GITR, IL10, TGF-B, OX40, TIM-1, and TIM-3 | inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Christophe MARIAT, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Nephrology Unit Hôpital Nord CHU de Saint-Etienne, Saint-Etienne, France

REFERENCES:
- [Background] Laville M, Alamartine E. Treatment options for IgA nephropathy in adults: a proposal for evidence-based strategy. Nephrol Dial Transplant. 2004 Aug;19(8):1947-51. doi: 10.1093/ndt/gfh309. Epub 2004 May 25. No abstract available. PMID 15161954
- [Background] Mariat C, Sanchez-Fueyo A, Alexopoulos SP, Kenny J, Strom TB, Zheng XX. Regulation of T cell dependent immune responses by TIM family members. Philos Trans R Soc Lond B Biol Sci. 2005 Sep 29;360(1461):1681-5. doi: 10.1098/rstb.2005.1706. PMID 16147532
- [Background] Mariat C Degauque N et al. TIM-1 strengthens Th-1 polarization and weakens CD4+CD25 T cells. Am J Transplant 6(suppl 2): 557, 2006